CLINICAL TRIAL: NCT02070861
Title: Non-invasive Volume Evaluation With Exhaled Carbon Dioxide and Pulse Contour Analysis (Nexfin)
Brief Title: Non-invasive Evaluation of Volume Status Using Exhaled Carbon Dioxide and Pulse Contour Analysis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Oslo University Hospital (Other)
Collaborators: The Norwegian Air Ambulance Foundation (Unknown)
Responsible Party: Principal Investigator, Ingrid Elise Hoff, MD, Oslo University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 2013/1605
Record Dates: First submitted 2014-02-23; First posted 2014-02-25 (Estimated); Last update posted 2018-04-17 (Actual); Status verified 2018-04

CONDITIONS: Changes in Cardiac Output
Keywords: Cardiac output; Exhaled CO2; Nexfin; Esophageal Doppler

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Comparing cardiac output changes (Experimental): Explore the relationship between changes in cardiac output measured with eosophagal Doppler, the volume-clamp-method and exhaled CO2 during ventricular pacing and passive leg raise.
  Measurements with the volume-clamp-method were aborted due to technological difficulties.
  Interventions: Other: Ventricular pacing and passive leg raise

INTERVENTIONS:
Other: Ventricular pacing and passive leg raise — Ventricular pacing and passive leg raise

SUMMARY:
The investigators hypothesize that changes in blood circulation can be reflected by exhaled CO2 provided CO2-production in the tissues and ventilation from the lungs are stable. The investigators want to explore changes in cardiac output (the amount of blood being pumped out of the heart each minute) in patients using different devices: an esophagus ultrasound device measuring cardiac output, a finger cuff measuring blood pressure and cardiac output, and exhaled carbondioxide in the patients' breath measured by the ventilator.

The investigators investigate patients after bypass surgery or heart valve replacement, and induce changes in cardiac output with passive leg raise or ventricular pacing.

DETAILED DESCRIPTION:
Measurements with the finger cuff (pulse contour analyses) were aborted due to technical difficulties.

ELIGIBILITY:
Inclusion Criteria:

* Persons 18 years or older scheduled to undergo arteriocoranary bypass surgery or aortic valve replacement.

Exclusion Criteria:

* Esophageal pathology, EF <40%

Ages: 18 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2014-04 (Actual); Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Changes in cardiac output | 5 Minutes

CONTACTS AND LOCATIONS:
Overall Officials: Leiv Arne Rosseland, MD, PhD, Study Chair — Oslo University Hospital
Locations (1):
- Oslo University Hospital, Ullevål, Oslo, Norway

IPD SHARING:
Plan to Share IPD: No
No plan to share individual participant data.

REFERENCES:
- [Derived] Hoff IE, Hoiseth LO, Kirkeboen KA, Landsverk SA. Volumetric and End-Tidal Capnography for the Detection of Cardiac Output Changes in Mechanically Ventilated Patients Early after Open Heart Surgery. Crit Care Res Pract. 2019 May 30;2019:6393649. doi: 10.1155/2019/6393649. eCollection 2019. PMID 31281675